CLINICAL TRIAL: NCT04040257
Title: Does a Team-based Approach Improve Knowledge and Judgment Performance in Electronic Fetal Monitoring?
Brief Title: A Team-based Approach to Improve Knowledge and Judgment Performance in Electronic Fetal Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000023716
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Electronic Fetal Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Performance (No Intervention): Each participant will first take the exam as an individual. After a delay of 3-6 months, participants will then be randomized to take the exam again either as an individual again (control group) or as a team (exposure group).
- Group Performance (Experimental): Each participant will first take the exam as an individual. After a delay of 3-6 months, participants will then be randomized to take the exam again either as an individual again (control group) or as a team (exposure group).
  Interventions: Behavioral: Team-based approach

INTERVENTIONS:
Behavioral: Team-based approach — Team-based participation in the The Perinatal Quality Foundation Fetal Monitoring Credentialing (PQF/FMC) exam.
  Arms: Group Performance

SUMMARY:
The primary objective of this study is to compare performance of nurses, midwives, and physicians working as individuals versus working as teams in electronic fetal monitoring (as assessed by differences in knowledge and judgment scores).

DETAILED DESCRIPTION:
Electronic fetal monitoring (EFM) has been used as a tool to evaluate fetal wellbeing in obstetrics for decades, with limited results with regard to improve fetal outcomes. There remains wide variation in the interpretation of fetal heart rate (FHR) tracings between different practitioners, which may explain the limited impact of this ubiquitous tool. The Perinatal Quality Foundation Fetal Monitoring Credentialing (PQF/FMC) exam was established to improve patient safety in obstetrical care by optimizing and standardizing the credentialing process for EFM.

The Fetal Monitoring Credentialing (FMC) test is a validated tool to assess the knowledge and judgment of test-takers based on script concordance theory, an approach to testing that allows assessment on real-life situations by comparing to the clinical reasoning of a panel of reference experts.

It is known that in clinical practice patients are cared for by teams of individuals (RN's, CNM, resident physicians and attendings). These individuals are all trained to approach a laboring patient from their own unique training. Even amongst experts in the field there is only moderate agreement on the interpretation of tracings with poor agreement on what constitutes a category III tracing. The absence of complete agreement in clinical practice creates differences in opinions of interpretation and agreement regarding next step in management for obstetric patients.

It is hypothesized that a team-based participation in the Perinatal Quality Foundation Fetal Monitoring Credentialing (PQF/FMC) exam will improve knowledge and judgment scores.

ELIGIBILITY:
Inclusion Criteria:

* Must be a registered nurse, certified midwife, physician (resident, attending, MFM and General OB/Gyn) and have full obstetric privileges to provide patient care at participating hospitals.

Exclusion Criteria:

* Any individual who does not meet inclusion criteria or is unable to participate in all exams at the designated time points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
The Perinatal Quality Foundation Fetal Monitoring Credentialing (PQF/FMC) Judgement | Up to 6 months
  The Perinatal Quality Foundation Fetal Monitoring Credentialing (PQF/FMC) exam measures judgement. The is exam is a 72 question computer based exam. There are 35 knowledge questions and 37 judgement questions. The scores for each section are reported as a percentage (maximum score = 100%). Knowledge and judgement questions have scores that are weighted based on exam key.
The Perinatal Quality Foundation Fetal Monitoring Credentialing (PQF/FMC) Knowledge | Up to 6 months
  The Perinatal Quality Foundation Fetal Monitoring Credentialing (PQF/FMC) exam measures knowledge. The is exam is a 72 question computer based exam. There are 35 knowledge questions and 37 judgement questions. The scores for each section are reported as a percentage (maximum score = 100%). Knowledge and judgement questions have scores that are weighted based on exam key.

CONTACTS AND LOCATIONS:
Overall Officials: Krista Mehlhaff, DO, Principal Investigator — Yale School of Medicine, Department of Obstetrics, Gynecology, & Reproductive Sciences
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No